CLINICAL TRIAL: NCT01081834
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin as Monotherapy in the Treatment of Subjects With Type 2 Diabetes Mellitus Inadequately Controlled With Diet and Exercise
Brief Title: The CANTATA-M (CANagliflozin Treatment and Trial Analysis - Monotherapy) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017011; 28431754DIA3005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Canagliflozin; Placebo; Hemoglobin A1c; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 52 weeks (Main Study) or 26 weeks only (High Glycemic Substudy).
  Interventions: Drug: Canagliflozin
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 52 weeks (Main Study) or 26 weeks only (High Glycemic Substudy).
  Interventions: Drug: Canagliflozin
- Placebo/Sitagliptin (Experimental): In the Main Study, each patient will receive matching placebo once daily for 26 weeks and will then switch from placebo to 100 mg of sitagliptin once daily until Week 52.
  Interventions: Drug: Placebo; Drug: Sitagliptin

INTERVENTIONS:
Drug: Canagliflozin — One 100 mg or 300 mg over-encapsulated tablet orally (by mouth) once daily for 52 weeks (Main Study) or 26 weeks (High Glycemic Substudy)
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Placebo — One matching placebo capsule orally once daily for 26 weeks (Main Study)
  Arms: Placebo/Sitagliptin
Drug: Sitagliptin — One 100 mg over-encapsulated tablet orally once daily beginning at Week 26 until Week 52 (Main Study)
  Arms: Placebo/Sitagliptin

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of 2 different doses of canagliflozin administered as monotherapy compared with placebo in patients with type 2 diabetes mellitus (T2DM) inadequately controlled with diet and exercise.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (study drug assigned by chance), double blind (neither the patient or the study doctor will know the name of the assigned treatment), parallel-group, 3 arm (patients will be assigned to 1 of 3 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of canagliflozin (100 mg and 300 mg) compared to placebo (a capsule that looks like all the other treatments but has no real medicine) in patients diagnosed with T2DM who are not achieving an adequate response from diet and exercise to control their diabetes. Approximately 450 patients with inadequate glycemic control with diet and exercise will receive once-daily treatment with canagliflozin 100 mg or 300 mg once daily for 52 weeks or 26 weeks of double-blind treatment with placebo followed by 26 weeks of sitagliptin 100 mg (sitagliptin is an antihyperglycemic agent that will allow patients randomized to the placebo group to improve glycemic control and remain in the study). Patients will participate in the study for approximately 60 to 68 weeks (referred to as the Main Study). The study will also include a High Glycemic Substudy in 50 to 100 patients with T2DM who have poorer glycemic control with diet and exercise. Patients in the substudy will be assigned to receive double-blind canagliflozin 100 mg or 300 mg for 26 weeks and the total duration of patient participatation in the substudy will be approximately 34 to 42 weeks. During treatment, if a patient's fasting blood sugar remains high despite treatment with study drug and reinforcement with diet and exercise, the patient will receive treatment with metformin (rescue therapy) consistent with local prescribing information. Study drug will be taken orally (by mouth) once daily before the first meal each day unless otherwise specified. Patients will take single blind placebo for 1 or 2 weeks (wks) before randomization to the Main Study or the High Glycemic Substudy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM
* Patients in the main study must have a Hemoglobin A1c (HbA1c) between >=7% and <=10% and a fasting plasma glucose (FPG) <270 mg/dL (15 mmol/L)
* Patients in the High Glycemic Cohort Substudy must have an HbA1c between >10% and <=12% and a FPG <=350 mg/dL (19.44 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, diabetes secondary to pancreatitis or pancreatectomy, or a severe hypoglycemic episode within 6 months before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (78):
- United States (24):
  - Phoenix, Arizona
  - Concord, California
  - Greenbrae, California
  - Los Angeles, California
  - Spring Valley, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Northglenn, Colorado
  - Springfield, Illinois
  - Evansville, Indiana
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Meridian, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - West Seneca, New York
  - Mooresville, North Carolina
  - Perryopolis, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Taylors, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Austria (3):
  - Horn
  - Salzburg
  - Vienna
- Colombia (2):
  - Barranquilla
  - Bogotá
- Estonia (3):
  - Pärnu
  - Tartu
  - Viljandi
- Guatemala City, Guatemala
- Reykjavik, Iceland
- India (3):
  - Bangalore
  - Hyderabad
  - Nagpur
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
  - Vilnius Lt
- Malaysia (2):
  - Kelantan
  - Kuala Lumpur
- Mexico (5):
  - Aguascalientes
  - Guadalajara
  - Mexico City
  - Monterrey
  - Zapopan
- Philippines (4):
  - Makati
  - Manila
  - Marikina City
  - Pasay
- Poland (3):
  - Katowice
  - Torun
  - Warsaw
- Puerto Rico (3):
  - Fajardo
  - Ponce
  - San Juan
- Romania (4):
  - Baia Mare
  - Brasov
  - Bucharest
  - Târgu Mureş
- South Africa (2):
  - Halfway
  - Pretoria
- South Korea (5):
  - Busan
  - Goyang-si
  - Jeonju
  - Seoul
  - Wŏnju
- Spain (4):
  - Alcalá de Henares
  - Elche
  - Girona
  - Pozuelo de Alarcón
- Sweden (4):
  - Gothenburg
  - Lund
  - Malmo
  - Skene

REFERENCES:
- [Derived] Davies MJ, Merton K, Vijapurkar U, Yee J, Qiu R. Efficacy and safety of canagliflozin in patients with type 2 diabetes based on history of cardiovascular disease or cardiovascular risk factors: a post hoc analysis of pooled data. Cardiovasc Diabetol. 2017 Mar 21;16(1):40. doi: 10.1186/s12933-017-0517-7. PMID 28327140
- [Derived] Pfeifer M, Townsend RR, Davies MJ, Vijapurkar U, Ren J. Effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on blood pressure and markers of arterial stiffness in patients with type 2 diabetes mellitus: a post hoc analysis. Cardiovasc Diabetol. 2017 Feb 27;16(1):29. doi: 10.1186/s12933-017-0511-0. PMID 28241822
- [Derived] Gilbert RE, Mende C, Vijapurkar U, Sha S, Davies MJ, Desai M. Effects of Canagliflozin on Serum Magnesium in Patients With Type 2 Diabetes Mellitus: A Post Hoc Analysis of Randomized Controlled Trials. Diabetes Ther. 2017 Apr;8(2):451-458. doi: 10.1007/s13300-017-0232-0. Epub 2017 Feb 14. PMID 28197834
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] John M, Cerdas S, Violante R, Deerochanawong C, Hassanein M, Slee A, Canovatchel W, Hamilton G. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus living in hot climates. Int J Clin Pract. 2016 Sep;70(9):775-85. doi: 10.1111/ijcp.12868. PMID 27600862
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Lavalle-Gonzalez FJ, Eliaschewitz FG, Cerdas S, Chacon Mdel P, Tong C, Alba M. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus from Latin America. Curr Med Res Opin. 2016;32(3):427-39. doi: 10.1185/03007995.2015.1121865. Epub 2016 Jan 14. PMID 26579834
- [Derived] Blonde L, Woo V, Mathieu C, Yee J, Vijapurkar U, Canovatchel W, Meininger G. Achievement of treatment goals with canagliflozin in patients with type 2 diabetes mellitus: a pooled analysis of randomized controlled trials. Curr Med Res Opin. 2015 Nov;31(11):1993-2000. doi: 10.1185/03007995.2015.1082991. Epub 2015 Sep 28. PMID 26373629
- [Derived] Gavin JR 3rd, Davies MJ, Davies M, Vijapurkar U, Alba M, Meininger G. The efficacy and safety of canagliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2015;31(9):1693-702. doi: 10.1185/03007995.2015.1067192. Epub 2015 Sep 4. PMID 26121561
- [Derived] Cefalu WT, Stenlof K, Leiter LA, Wilding JP, Blonde L, Polidori D, Xie J, Sullivan D, Usiskin K, Canovatchel W, Meininger G. Effects of canagliflozin on body weight and relationship to HbA1c and blood pressure changes in patients with type 2 diabetes. Diabetologia. 2015 Jun;58(6):1183-7. doi: 10.1007/s00125-015-3547-2. Epub 2015 Mar 27. PMID 25813214
- [Derived] Weir MR, Januszewicz A, Gilbert RE, Vijapurkar U, Kline I, Fung A, Meininger G. Effect of canagliflozin on blood pressure and adverse events related to osmotic diuresis and reduced intravascular volume in patients with type 2 diabetes mellitus. J Clin Hypertens (Greenwich). 2014 Dec;16(12):875-82. doi: 10.1111/jch.12425. Epub 2014 Oct 20. PMID 25329038
- [Derived] Usiskin K, Kline I, Fung A, Mayer C, Meininger G. Safety and tolerability of canagliflozin in patients with type 2 diabetes mellitus: pooled analysis of phase 3 study results. Postgrad Med. 2014 May;126(3):16-34. doi: 10.3810/pgm.2014.05.2753. PMID 24918789
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Sinclair A, Bode B, Harris S, Vijapurkar U, Mayer C, Fung A, Shaw W, Usiskin K, Desai M, Meininger G. Efficacy and safety of canagliflozin compared with placebo in older patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. BMC Endocr Disord. 2014 Apr 18;14:37. doi: 10.1186/1472-6823-14-37. PMID 24742013
- [Derived] Polidori D, Mari A, Ferrannini E. Canagliflozin, a sodium glucose co-transporter 2 inhibitor, improves model-based indices of beta cell function in patients with type 2 diabetes. Diabetologia. 2014 May;57(5):891-901. doi: 10.1007/s00125-014-3196-x. Epub 2014 Mar 1. PMID 24585202
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339
- [Derived] Stenlof K, Cefalu WT, Kim KA, Jodar E, Alba M, Edwards R, Tong C, Canovatchel W, Meininger G. Long-term efficacy and safety of canagliflozin monotherapy in patients with type 2 diabetes inadequately controlled with diet and exercise: findings from the 52-week CANTATA-M study. Curr Med Res Opin. 2014 Feb;30(2):163-75. doi: 10.1185/03007995.2013.850066. Epub 2013 Oct 28. PMID 24073995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus inadequately controlled with diet and exercise. The study was conducted between 08 February 2010 and 18 August 2011 and recruited patients from 90 study centers in 17 countries worldwide.
Pre-assignment Details: 678 patients were enrolled into the study; 587 patients in the main study and 91 patients in the high glycemic substudy. 584 patients in the main study and all 91 patients in the high glycemic substudy received at least one dose of study drug and were included in the modified intent-to-treat (mITT) analyses sets and the safety analyses sets.
Groups:
- Main Study: Placebo/Sitagliptin: In the Main Study, each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52.
- Main Study: Canagliflozin 100 mg: In the Main Study, each patient received 100 mg of canagliflozin once daily for 52 weeks.
- Main Study: Canagliflozin 300 mg: In the Main Study, each patient received 300 mg of canagliflozin once daily for 52 weeks.
- High Glycemic Substudy: Canagliflozin 100 mg: In the High Glycemic Substudy, each patient received 100 mg of canagliflozin once daily for 26 weeks only. No patients received treatment during the period Week 26 to Week 52.
- High Glycemic Substudy: Canagliflozin 300 mg: In the High Glycemic Substudy, each patient received 300 mg of canagliflozin once daily for 26 weeks only. No patients received treatment during the period Week 26 to Week 52.
Period: Core Period: Baseline to Week 26
Arm/Group | Main Study: Placebo/Sitagliptin | Main Study: Canagliflozin 100 mg | Main Study: Canagliflozin 300 mg | High Glycemic Substudy: Canagliflozin 100 mg | High Glycemic Substudy: Canagliflozin 300 mg
Started | 192 | 195 | 197 | 47 | 44
Completed | 160 | 172 | 175 | 40 | 40
Not Completed | 32 | 23 | 22 | 7 | 4
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 5 | 3 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 5 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 15 | 3 | 9 | 3 | 1
Not completed — Noncompliance with study drug | 3 | 4 | 2 | 2 | 0
Not completed — Unable to take rescue therapy | 1 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 4 | 3 | 1 | 0
Not completed — Lack of efficacy on rescue therapy | 3 | 1 | 0 | 0 | 0
Period: Extension Period: Week 26 to Week 52
Arm/Group | Main Study: Placebo/Sitagliptin | Main Study: Canagliflozin 100 mg | Main Study: Canagliflozin 300 mg | High Glycemic Substudy: Canagliflozin 100 mg | High Glycemic Substudy: Canagliflozin 300 mg
Started | 155 (5 pts discontinued on last day of core: lack of efficacy on rescue (2), not specified (NS) (3).) | 170 (2 pts discontinued on last day of core: adverse event (AE) (1), protocol violation (PV) (1).) | 170 (5 pts discontinued last day of core: AE (1), lost f/u (1), PV (1), NS (1), physician decision (1).) | 0 (The treatment duration for the High Glycemic Substudy was 26 weeks only.) | 0 (The treatment duration for the High Glycemic Substudy was 26 weeks only.)
Completed | 135 | 152 | 165 | 0 | 0
Not Completed | 20 | 18 | 5 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0
Not completed — Unable to take rescue therapy | 1 | 0 | 1 | 0 | 0
Not completed — Creatinine or eGFR withdrawal criteria | 1 | 4 | 0 | 0 | 0
Not completed — Other | 4 | 5 | 4 | 0 | 0
Not completed — Lack of efficacy on rescue therapy | 7 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Glycemic Substudy: Canagliflozin 100 mg: In the High Glycemic Substudy, each patient received 100 mg of canagliflozin once daily for 26 weeks.
- High Glycemic Substudy: Canagliflozin 300 mg: In the High Glycemic Substudy, each patient received 300 mg of canagliflozin once daily for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Main Study: Placebo/Sitagliptin | Main Study: Canagliflozin 100 mg | Main Study: Canagliflozin 300 mg | High Glycemic Substudy: Canagliflozin 100 mg | High Glycemic Substudy: Canagliflozin 300 mg | Total
Number analyzed (Participants) | 192 | 195 | 197 | 47 | 44 | 675
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 150 | 156 | 160 | 42 | 41 | 549
  >=65 years | 42 | 39 | 37 | 5 | 3 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.88) | 55.1 (10.83) | 55.3 (10.17) | 49.7 (11.12) | 48.8 (10.92) | 54.5 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 114 | 108 | 24 | 25 | 375
  Male | 88 | 81 | 89 | 23 | 19 | 300
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 1 | 2 | 1 | 0 | 0 | 4
  COLOMBIA | 8 | 8 | 6 | 3 | 0 | 25
  ESTONIA | 6 | 5 | 5 | 0 | 0 | 16
  GUATEMALA | 10 | 10 | 13 | 9 | 10 | 52
  ICELAND | 4 | 4 | 8 | 2 | 2 | 20
  INDIA | 8 | 11 | 8 | 5 | 2 | 34
  LITHUANIA | 17 | 10 | 12 | 2 | 1 | 42
  MALAYSIA | 6 | 2 | 7 | 1 | 0 | 16
  MEXICO | 19 | 23 | 19 | 2 | 2 | 65
  PHILIPPINES | 3 | 4 | 6 | 4 | 4 | 21
  POLAND | 1 | 4 | 3 | 0 | 0 | 8
  ROMANIA | 20 | 16 | 18 | 2 | 4 | 60
  SOUTH AFRICA | 9 | 6 | 11 | 1 | 2 | 29
  SOUTH KOREA | 10 | 8 | 7 | 1 | 1 | 27
  SPAIN | 3 | 2 | 3 | 0 | 0 | 8
  SWEDEN | 11 | 18 | 18 | 0 | 1 | 48
  UNITED STATES | 56 | 62 | 52 | 15 | 15 | 200

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 26 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Placebo: In the Main Study, each patient recieved matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52.
- Canagliflozin 100 mg: In the Main Study, each patient received 100 mg of canagliflozin once daily for 52 weeks.
- Canagliflozin 300 mg: In the Main Study, each pateint received 300 mg of canagliflozin once daily for 52 weeks.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 189 | 191 | 194
Percent | 0.14 (0.065) | -0.77 (0.065) | -1.03 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.91, 95% CI 2-sided [-1.088 to -0.729], Standard Error of Mean 0.091
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.16, 95% CI 2-sided [-1.342 to -0.985], Standard Error of Mean 0.091

2. Primary Outcome: Change in HbA1c From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Placebo: In the High Glycemic Substudy, no patients received placebo.
- Canagliflozin 100 mg: In the High Glycemic Substudy, each patient received 100 mg of canagliflozin once daily for 26 weeks.
- Canagliflozin 300 mg: In the High Glycemic Substudy, each pateint received 300 mg of canagliflozin once daily for 26 weeks.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 46 | 43
Percent |  | -2.13 (0.220) | -2.56 (0.227)

3. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26 (Main Study)
Description: The table below shows the percentage of patients with HbA1c <7% at Week 26. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 189 | 191 | 194
Percentage of patients | 20.6 | 44.5 | 62.4
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.34, 95% CI 2-sided [3.10 to 9.23]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.61, 95% CI 2-sided [8.14 to 26.25]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Placebo: In the Main Study, each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 184 | 188 | 192
mg/dL | 8.33 (2.448) | -27.2 (2.412) | -35.0 (2.391)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -35.5, 95% CI 2-sided [-42.22 to -28.78], Standard Error of Mean 3.420
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -43.4, 95% CI 2-sided [-50.06 to -36.69], Standard Error of Mean 3.402

5. Secondary Outcome: Change in 2-hour Post-prandial Glucose From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean change in 2-hour post-prandial glucose from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 126 | 154 | 157
mg/dL | 5.19 (4.204) | -42.9 (3.763) | -58.8 (3.741)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -49.1, 95% CI 2-sided [-59.12 to -36.99], Standard Error of Mean 5.629
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -64.0, 95% CI 2-sided [-75.02 to -52.94], Standard Error of Mean 5.616

6. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 190 | 192 | 194
Percent change | -0.6 (0.2) | -2.8 (0.2) | -3.9 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.2, 95% CI 2-sided [-2.9 to -1.6], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -3.3, 95% CI 2-sided [-4.0 to -2.6], Standard Error of Mean 0.3

7. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 190 | 192 | 195
mmHg | 0.38 (0.780) | -3.34 (0.775) | -5.04 (0.769)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -3.71, 95% CI 2-sided [-5.860 to -1.568], Standard Error of Mean 1.093
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -5.42, 95% CI 2-sided [-7.556 to -3.280], Standard Error of Mean 1.088

8. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean percent change in triglycerides from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 171 | 183 | 183
Percent change | 7.8 (3.5) | 2.5 (3.3) | -2.4 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.267, ANCOVA; Least-Squares Mean Difference = -5.3, 95% CI 2-sided [-14.8 to 4.1], Standard Error of Mean 4.8
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.034, ANCOVA; Least-Squares Mean Difference = -10.2, 95% CI 2-sided [-19.6 to -0.8], Standard Error of Mean 4.8

9. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26 (Main Study)
Description: The table below shows the least-squares (LS) mean percent change in HDL-C from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 170 | 182 | 183
Percent change | 4.4 (1.4) | 11.2 (1.4) | 10.5 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 6.7, 95% CI 2-sided [2.9 to 10.6], Standard Error of Mean 1.9
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; Least-Squares Mean Difference = 6.0, 95% CI 2-sided [2.2 to 9.9], Standard Error of Mean 1.9

10. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26 (High Glycemic Substudy)
Description: The table below shows the percentage of patients with HbA1c <7% at Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 46 | 43
Percentage of patients |  | 17.4 | 11.6

11. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 45 | 43
mg/dL |  | -81.7 (6.459) | -86.3 (6.553)

12. Secondary Outcome: Change in 2-hour Post-prandial Glucose From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares (LS) mean change in 2-hour post-prandial glucose from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 30 | 34
mg/dL |  | -118 (10.179) | -126 (9.437)

13. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 46 | 43
Percent change |  | -3.0 (0.6) | -3.8 (0.6)

14. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 46 | 43
mmHg |  | -4.47 (1.754) | -4.97 (1.800)

15. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares mean percent change in triglycerides from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 44 | 43
Percent change |  | -0.6 (7.4) | -12.7 (7.5)

16. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26 (High Glycemic Substudy)
Description: The table below shows the least-squares mean percent change in HDL-C from Baseline to Week 26 for each treatment group in patients randomized to the High Glycemic Substudy.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 0 | 44 | 43
Percent change |  | 2.4 (2.9) | 10.8 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 52 weeks.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Groups:
- Main Study (Baseline to Week 26): Placebo: Each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52. Data are presented for Baseline to Week 26.
- Main Study (Baseline to Week 26): Cana 100 mg: Each patient received 100 mg of canagliflozin (Cana) once daily for 52 weeks. Data are presented for Baseline to Week 26.
- Main Study (Baseline to Week 26): Cana 300 mg: Each patient received 300 mg of canagliflozin (Cana) once daily for 52 weeks. Data are presented for Baseline to Week 26.
- Main Study (Baseline to Week 52): Placebo/Sitagliptin: Each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52. Data are presented for Baseline to Week 52.
- Main Study (Baseline to Week 52): Cana 100 mg: Each patient received 100 mg of canagliflozin (Cana) once daily for 52 weeks. Data are presented for Baseline to Week 52.
- Main Study (Baseline to Week 52): Cana 300 mg: Each patient received 300 mg of canagliflozin (Cana) once daily for 52 weeks. Data are presented for Baseline to Week 52.
- High Glycemic Substudy (Baseline to Week 26): Cana 100 mg: Each patient received 100 mg of canagliflozin (Cana) once daily for 26 weeks. Data are only available for Baseline to Week 26.
- High Glycemic Substudy (Baseline to Week 26): Cana 300 mg: Each patient received 300 mg of canagliflozin (Cana) once daily for 26 weeks. Data are only available for Baseline to Week 26.
Arm/Group | Main Study (Baseline to Week 26): Placebo | Main Study (Baseline to Week 26): Cana 100 mg | Main Study (Baseline to Week 26): Cana 300 mg | Main Study (Baseline to Week 52): Placebo/Sitagliptin | Main Study (Baseline to Week 52): Cana 100 mg | Main Study (Baseline to Week 52): Cana 300 mg | High Glycemic Substudy (Baseline to Week 26): Cana 100 mg | High Glycemic Substudy (Baseline to Week 26): Cana 300 mg
Serious Adverse Events (participants affected / at risk) | 4/192 | 8/195 | 2/197 | 11/192 | 11/195 | 5/197 | 0/47 | 1/44
Other Adverse Events (participants affected / at risk) | 38/192 | 39/195 | 51/197 | 63/192 | 54/195 | 69/197 | 6/47 | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study (Baseline to Week 26): Placebo (N=192) | Main Study (Baseline to Week 26): Cana 100 mg (N=195) | Main Study (Baseline to Week 26): Cana 300 mg (N=197) | Main Study (Baseline to Week 52): Placebo/Sitagliptin (N=192) | Main Study (Baseline to Week 52): Cana 100 mg (N=195) | Main Study (Baseline to Week 52): Cana 300 mg (N=197) | High Glycemic Substudy (Baseline to Week 26): Cana 100 mg (N=47) | High Glycemic Substudy (Baseline to Week 26): Cana 300 mg (N=44)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial prostatitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral pericarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study (Baseline to Week 26): Placebo (N=192) | Main Study (Baseline to Week 26): Cana 100 mg (N=195) | Main Study (Baseline to Week 26): Cana 300 mg (N=197) | Main Study (Baseline to Week 52): Placebo/Sitagliptin (N=192) | Main Study (Baseline to Week 52): Cana 100 mg (N=195) | Main Study (Baseline to Week 52): Cana 300 mg (N=197) | High Glycemic Substudy (Baseline to Week 26): Cana 100 mg (N=47) | High Glycemic Substudy (Baseline to Week 26): Cana 300 mg (N=44)
Nasopharyngitis (Infections and infestations) | 10 | 10 | 16 | 15 | 14 | 20 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 11 | 7 | 9 | 18 | 8 | 14 | 0 | 0
Urinary tract infection (Infections and infestations) | 8 | 14 | 9 | 11 | 16 | 12 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 12 | 9 | 5 | 15 | 0 | 0
Headache (Nervous system disorders) | 7 | 14 | 12 | 12 | 19 | 17 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 7 | 12 | 8 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 13 | 10 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.